CLINICAL TRIAL: NCT02585076
Title: A National, Multicenter, Non-interventional, Crosssectional Study for the Determination of the pREvalence of Non-valvular Atrial FIbrillation Among patieNts Diagnosed With Hypertension Attending HEllenic Hypertension Centers
Brief Title: A Cross-sectional Study for the Determination of the Prevalence of Non-valvular Atrial Fibrillation Among Patients Diagnosed With Hypertension
Acronym: REFINE HT
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 18311
Record Dates: First submitted 2015-10-20; First posted 2015-10-23 (Estimated); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Hypertension; Atrial Fibrillation
Keywords: Stroke prevention; Risk assessment
MeSH Terms: conditions — Hypertension; Atrial Fibrillation | interventions — Standard of Care

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cohort 1: Patients aged 60 years or older regardless of gender and race with a documented diagnosis of hypertension will be enrolled into this study after the decision for electrocardiographic screening for AF has been made by the investigator
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Standard of care — As prescribed by treated physician

SUMMARY:
Arterial hypertension has been recognized as a major causal factor for atrial fibrillation (AF), the most common sustained cardiac arrhythmia. In light of its worldwide increasing prevalence and incidence and the accompanied increase in the risk of stroke, thromboembolic events and mortality, AF has emerged as a global healthcare problem.

Early diagnosis of AF, prior to the occurrence of complications is a recognized priority for the prevention of strokes. Once diagnosed, anticoagulant therapy is the cornerstone in the management of the risk of stroke in AF patients. The 2012 ESC Guidelines recommend the use of a risk factor-based approach to stroke risk stratification for AF patients.

This study aims towards gaining real-world data on the prevalence of non-valvular atrial fibrillation (NVAF) among hypertensives in Greece. The rate of ESC guideline-adherent antithrombotic therapy on the basis of stroke and bleeding risk assessments, and factors influencing treatment decision-making will be assessed as well in patients diagnosed with the arrhythmia.

Finally, potential differences in the NVAF prevalence in adequately and inadequately controlled hypertensives will be documented.

ELIGIBILITY:
Inclusion Criteria:

* Female and male outpatients aged 60 years and older
* Patients having being diagnosed with arterial hypertension
* For patients without a history of AF diagnosis, the decision to perform electrocardiography testing, either standard 12-lead ECG or ambulatory ECG, at the study visit has been made as per the investigator's routine practice
* Patients with available medical records
* Written signed and dated informed consent

Exclusion Criteria

* Presence of any condition/circumstance which in the opinion of the investigator would make the patient unfit to participate in the study or would compromise the quality of the study data (e.g., non-native speaker or patient who does not understand the local language unless reliable interpreter services are available; failure to cooperate due to major psychiatric disturbances, dementia, or substance use disorder)
* Patients currently participating in any investigational program with interventions outside of routine clinical practice or who have received any investigational product within 1 month or 5 half-lives of the investigational agent (whichever is longer) prior to enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be carried out by hypertension specialists practicing in the hospital-based outpatient healthcare sector, among the network of the European Society of Hypertension (ESH) Hypertension Excellence Centers
Sampling Method: Probability Sample
Enrollment: 1119 (Actual)
Dates: Start 2015-11-04 (Actual); Primary Completion 2016-02-29 (Actual); Study Completion 2016-05-30 (Actual)

PRIMARY OUTCOMES:
Frequency of non-valvular atrial fibrillation (NAVF) among hypertensive outpatients | At enrollment

SECONDARY OUTCOMES:
Proportion of NVAF patients for whom the HAS-BLED score has been estimated by the physicians as part of the decision for antithrombotic treatment | At enrollment
  HAS-BLED: Hypertension, Abnormal renal/liver function, Stroke, Bleeding history or predisposition, Labile INR, Elderly, Drugs/alcohol concomitantly
Frequency of oral anticoagulation therapy among the study population diagnosed with NVAF | At enrollment
Proportion of untreated patients among the study population diagnosed with NVAF | At enrollment
Proportion of antiplatelet therapy treated patients among the study population diagnosed with NVAF | At enrollment
CHADS2 scores | At enrollment
  CHADS2 : Congestive heart failure, Hypertension, Age 75 years or older, Diabetes mellitus and prior Stroke or transient ischemic attack (doubled)
CHA2DS2-VASc scores | At enrollment
  CHA2DS2-VASc: Congestive heart failure, Hypertension, Age 75 years or older (doubled), Diabetes mellitus, previous Stroke/transient ischemic attack (doubled), Vascular disease, Age 65-74 years and Sex category
Degree of agreement between the proportions of patients classified at intermediate and high stroke risk according to the two risk stratification systems | At enrollment
CHA2DS2-VASc score in hypertensives without NVAF | At enrollment
Correlation of the CHA2DS2-VASc-assessed risk with the average annual stroke risk as calculated by the Framingham stroke risk scoring system in hypertensives without NVAF | At enrollment
  A Poisson regression model or negative binomial model will be applied in order to examine the potential association of the Framingham stroke risk score with the CHA2DS2-VASc score
CHA2DS2-VASc score in hypertensives without AF | At enrollment
Correlation of the CHA2DS2-VASc-assessed risk with the average annual AF risk as calculated by the Framingham AF risk scoring system in hypertensives without AF | At enrollment
  A Poisson regression model or negative binomial model will be applied in order to examine the potential association of the Framingham AF risk score with the CHA2DS2-VASc score
Frequency of NVAF among the subpopulations of hypertensives adequately versus those inadequately controlled according to the physicians' medical judgement | At enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Greece